CLINICAL TRIAL: NCT02401217
Title: Tolerance of Healthy Infants Fed Infant Formulas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: AL12
Record Dates: First submitted 2015-03-16; First posted 2015-03-27 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Gastrointestinal Tolerance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Phase 1-Arm 1 Infant Formula (Experimental): Milk-based infant formula manufactured by an alternative method. Non-commercially available formula. To be fed ad libitum.
  Interventions: Other: Phase 1- Arm 1 Infant Formula
- Phase 2- Arm 2 Infant Formula (Active Comparator): Milk-based infant formula using current manufacturing and ingredients. Non-commercially available formula. To be fed ad libitum.
  Interventions: Other: Phase 2- Arm 2 Infant Formula
- Phase 2- Arm 3 Infant Formula (Experimental): Milk-based infant formula using a new protein. Non-commercially available formula. To be fed ad libitum.
  Interventions: Other: Phase 2- Arm 3 Infant Formula

INTERVENTIONS:
Other: Phase 1- Arm 1 Infant Formula — Powder infant formula
  Arms: Phase 1-Arm 1 Infant Formula
Other: Phase 2- Arm 2 Infant Formula — Powder infant formula
  Arms: Phase 2- Arm 2 Infant Formula
Other: Phase 2- Arm 3 Infant Formula — Powder infant formula
  Arms: Phase 2- Arm 3 Infant Formula

SUMMARY:
The primary objective of this study is to assess the comparative gastrointestinal tolerance of normal term infants to two experimental milk-based powdered formulas compared with a standard milk-based powdered formula.

ELIGIBILITY:
Inclusion Criteria:

* Singleton from a full term birth with a gestational age of 37-42 weeks.
* Birth weight was > 2490 g (~5 lbs 8 oz).
* Age between 0 and 30 days at enrollment.
* Agreement to discontinue the use of medications (including over the counter [OTC], such as Mylicon® for gas), home remedies, herbal preparations or rehydration fluids that might affect GI tolerance for the duration of the study.
* Intention to feed the infant the study product as the sole source of nutrition for the duration of the study.
* Intention not to administer vitamin (other than Vitamin D) or mineral supplements, solid foods or juices to their infant from enrollment through the duration of the study.
* Voluntarily signed and dated an informed consent form (ICF) approved by an Independent Ethics Committee/Institutional Review Board (IEC/IRB) and provided Health Insurance Portability and Accountability Act (HIPAA) (or other applicable privacy regulation) authorization prior to any participation in the study.

Exclusion Criteria:

* An adverse maternal, fetal or infant medical history that is thought by the investigator to have potential for effects on tolerance, growth, and/or development.
* Infant treated with antibiotics.
* Participation in another study that has not been approved as a concomitant study by AN.

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Stool consistency measured by Mean Rank Stool Consistency (MRSC) using parent reported diaries | Change from Study Day 1 to Study Day 15
  MRSC will be calculated from data recorded on daily stool records during the study. Stool consistencies will be assigned the following: 1=watery, 2=loose/mushy, 3=soft, 4=formed, 5=hard.

SECONDARY OUTCOMES:
Mean Percentage of stools representing each stool consistency and color using parent reported diaries | Change from Study Day 1 to Study Day 15
  Mean percentage of each recorded stool consistency (watery, loose/mushy, soft, formed, hard) and stool color (yellow, brown, green, black) will be calculated for each infant and then used to calculate for each group from daily data recorded on daily stool records during the study.
Mean predominant stool consistency and color measured using parent reported diaries | Change from Study Day 1 to Study Day 15
  Mean predominant stool consistency and color for each infant calculated from data recorded on daily stool records during the study will be used to calculate the mean predominant stool consistency and color for each group.
Average number of stools per day measured using parent reported diaries | Change from Study Day 1 to Study Day 15
  Average number of stools/day will be calculated for each group from data recorded on daily stool records during the study.
Mean percentages of feedings associated with spit-up and/or vomit measured using parent reported diaries. | Change from Study Day 1 to Study Day 15
  Mean percentages of feedings associated with spit-up and/or vomiting will be calculated for each group from data recorded on daily formula intake records during the study.
Parental responses to Formula Satisfaction and Infant Feeding and Stool Patterns Questionnaires | Change from Study Day 1 to Study Day 15
  Parental responses to individual question on the Formula Satisfaction Questionnaire will be calculated from data recorded on the questionnaire at Study Day 15
Parental assessment of infant feeding and stool patterns measured by the Infant Feeding and Stool Patterns Questionnaire. | Change from Study Day 1 to Study Day 15
  Parental responses to individual question on the Feeding and Stool Patterns Questionnaire will be calculated from data recorded on the questionnaire at Study Day 15.

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Borschel, PhD, RD, Study Chair — Abbott Nutrition
Locations (6):
- United States (6):
  - W.O.M.B Watching Over Mothers and Babies, Tucson, Arizona
  - SCORE Physician Alliance LLC, St. Petersburg, Florida
  - White Oak Family Physicians DBA/Asheboro Research Associates, Asheboro, North Carolina
  - Institute of Clinical Research, LLC, Mayfield Heights, Ohio
  - The Cleveland Pediatric Research Center, LLC, Middleburg Heights, Ohio
  - Tanner Memorial Clinic, Layton, Utah